CLINICAL TRIAL: NCT06736236
Title: Effects of Inspiratory Muscle Warm-up on Diffusion Capacity for Carbon Monoxide, Cardiorespiratory, Perceptual and Performance Outcomes During High-intensity Exercise in Elite Athletes from Different Disciplines: a Randomized, Placebo-controlled, Double-blind and Crossover Study
Brief Title: The Effect of Respiratory Muscle Warm-up on Pulmonary Diffusion Capacity in Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Karaduman (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor-Investigator, Emre Karaduman, Research Asistant, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PYO.YDS.1901.22.002
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healty Male Volunteers; Athlete
Keywords: inspiratory muscle warm-up; warm-up; DLCO

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Other): Participants only performed a general warm-up exercise.
  Interventions: Other: General warm-up (Control)
- IMW %15 (Placebo) (Placebo Comparator): In addition to the general warm-up, the participants performed IMW at 15% resistance intensity.
  Interventions: Other: Inspiratory muscle warm-up placebo (IMW %15)
- IWM %40 (Experimental) (Experimental): In addition to the general warm-up, participants performed IMW at 40% resistance intensity.
  Interventions: Other: Inspiratory muscle warm-up

INTERVENTIONS:
Other: Inspiratory muscle warm-up — This study will use a respiratory muscle warm-up protocol set at 40% of the maximal inspiratory pressure (MIP) using the POWERbreath® device, as this intensity has been shown to optimally stimulate respiratory muscles. The protocol involves two sets of 30 breaths with a 60-second rest between sets, performed with participants sitting and using a nose clip. Participants will be trained in this technique during the familiarization session and monitored throughout the tests to ensure proper execution.
  Other Names: Respiratory muscle warm-up
  Arms: IWM %40 (Experimental)
Other: General warm-up (Control) — The general warm-up (Control) protocol will include exercises such as running and dynamic, active, and passive movements tailored to the diverse sports disciplines in the study. These movements will follow the principles of elevation, activation, and mobilization, focusing on increasing mobility from the arms and shoulders to the lower back and legs. Each session will involve demonstrations emphasizing proper technique and speed, with participants completing a consistent number of repetitions. Researchers will monitor participants closely to ensure correct form and execution throughout the intervention.
  Arms: Control
Other: Inspiratory muscle warm-up placebo (IMW %15) — The respiratory muscle warm-up protocol will be conducted at 15% of maximal inspiratory pressure (MIP) using the POWERbreath® device. This placebo protocol will involve two sets of 30 breaths, separated by a 60-second rest, with participants seated and wearing a nose clip. Training for the technique will occur during a familiarization session, and participants will be observed during tests to ensure proper execution. The purpose of this protocol is to serve as a placebo, masking the actual aim of the study to enhance data reliability.
  Arms: IMW %15 (Placebo)

SUMMARY:
Several studies suggest that inspiratory muscle warm-up (IMW) could potentially affect exercise performance; however, its mechanistic basis is still unclear. The aim of this study was to examine the effect of IMW on lung diffusing capacity for carbon monoxide, cardiorespiratory, perceptual and performance outcomes in elite athletes from different disciplines.

The aim of this study is to evaluate the effects of IMW on diffusion capacity for carbon monoxide, cardiorespiratory, perceptual and performance outcomes during high-intensity exercise in elite athletes from different disciplines. The study will be conducted using a randomized, placebo-controlled, double-blind and crossover study experimental design involving 35 athletes from various sports disciplines, including endurance, strength, skill-based, and mixed disciplines.

Participants will attend the laboratory on four separate occasions. During the first visit, they will be informed about the study and familiarized with the application and measurement procedures. In the second visit, a general warm-up will be performed. During the third and fourth visits, IMW (IMW40% or IMW placebo) protocols will be applied in addition to the general warm-up. Measurements of DLCO, pulmonary function tests, respiratory muscle strength, and gas analysis during maximal aerobic exercise will be collected both before and after the warm-up protocols.

DETAILED DESCRIPTION:
A. STUDY DESING This study will employ a placebo-controlled, randomized, crossover, and double-blind research design to evaluate the effects of three warm-up conditions: Control, Placebo 15%, and IMW 40%. Athletes will be randomly assigned to the conditions using a crossover approach, ensuring that all participants will experience each protocol on separate days.

The warm-up protocols will include:

General Warm-up (Control): A standard warm-up without resistance. IMW 40%: A general warm-up combined with respiratory muscle exercise at 40% resistance.

Placebo 15%: A general warm-up combined with placebo respiratory muscle exercise at 15% resistance.

Blinding will be maintained for both participants and researchers. Participants will be informed that the study aims to investigate various warm-up types, while the true purpose will remain concealed. This design will ensure reliability and minimize bias in the data to be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-24 years.
* A training history of at least six years.
* Regular training frequency of at least four sessions per week.

Exclusion Criteria:

* History of smoking.
* History of physical disability or acute respiratory or cardiovascular disease within the past three months.
* Diagnosis of SARS-CoV-2 within the past three months.
* Pulmonary function measurements outside the normal clinical range (≤ 80%).

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Lung Carbon Monoxide Diffusion Capacity (DLCO) | Pre intervention and immediately post intervention
  DLCO will be measured using the single breath-hold method with a Quark PFT gas analyzer, following ATS/ERS standards. Each test involves inhalation of a gas mixture (0.3% CO, 0.3% CH4, and dry air), breath-holding for 10±2 seconds, and exhalation. Subjects will perform two DLCO tests at baseline, after warm-up protocols, and after VO2max testing during each laboratory visit.
Pulmonary Functions | Pre intervention and immediately post intervention
  Pulmonary function will be assessed using the Quark PFT device according to ATS/ERS guidelines. Respiratory function will be assessed using forced, slow, and maximal voluntary maneuvers. Subjects will perform specific maneuvers for each parameter while seated, with disposable mouthpieces and a nose clip to ensure accurate recordings.
Respiratory Muscle Strength | Pre intervention and immediately post intervention
  Respiratory muscle strength will be measured using the Pony FX MIP/MEP device following ERS guidelines. For maximal inspiratory pressure (MIP), subjects will exhale maximally, followed by a maximal inspiration against a closed valve. At least three trials with less than 5% variability will be averaged to determine the final values.
Respiratory Muscle Strength | Pre intervention and immediately post intervention
  Respiratory muscle strength will be measured using the Pony FX MIP/MEP device following ERS guidelines. For maximal expiratory pressure (MEP), subjects will inhale maximally, followed by a maximal expiration against a closed valve. At least three trials with less than 5% variability will be averaged to determine the final values.
Bicycle ergometer and Maximal Aerobic Capacity (VO2max) | Pre intervention and immediately post intervention
  The test will begin at a workload of 50 (Watt) and will progress by increasing the workload by 25 (Watt) every two minutes. Throughout the test, the pedaling speed (rhythm) will be continuously monitored on the bicycle display, and participants will be instructed to maintain a steady pace within an average range of ≥60 (±5) rpm. Despite strong verbal encouragement provided during the test, it will be terminated if a participant spends more than 10 seconds below the 55 rpm pedal rhythm and decides they cannot continue further (voluntary exhaustion). After completing the test, participants will continue pedaling at a workload of 20 (Watt) for approximately 2 minutes for active recovery. Each test will be initiated in accordance with the workload optimization and adjustments to bike fit (saddle, handlebar height, and position) performed during the first visit.
  Cardiopulmonary data will be obtained using a breath-by-breath Quark CPET metabolic system (Mixing chamber system) (COSMED, Alban

IPD SHARING:
Plan to Share IPD: Undecided